CLINICAL TRIAL: NCT04659681
Title: Role of Lung Ultrasonography in Detecting Extravascular Lung Water in Major Oncosurgeries
Acronym: LUS EVLW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Primary Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RajivGCIRC LUS
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Extravascular Lung Water
Keywords: Lung Ultrasonography Extravascular Lung Water Plethysmography variability Index

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant was masked about Group it belonged
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI Guided Fluid Therapy (Active Comparator): Patients will receive PVI guided fluids during surgery PVI to be maintained below 12% if PVI >12 then colloid bolus 200ml will be given. Lung Ultrasonography will be performed post-intubation as baseline and at the end of surgery before extubation in 4 Lung zones in both lungs to measure total number of B-lines.
  Interventions: Diagnostic Test: PVI Guided fluid management during surgery for (PVI<12) colloid bolus will be given .
- CVP Guided Fluid Therapy (Active Comparator): Patients will receive Standard CVP Guided Fluids , CVP maintained between 10-16 cms H20 , if CVP< 10 then colloid bolus 200ml will be given. Lung Ultrasonography will be performed post-intubation as baseline and at the end of surgery before extubation in 4 zones in both lungs to measure total number of B-lines.
  Interventions: Diagnostic Test: CVP Guided Fluid management during surgery for CVP<10 cms H2O colloid bolus will be given

INTERVENTIONS:
Diagnostic Test: PVI Guided fluid management during surgery for (PVI<12) colloid bolus will be given . — PVI probe attached to finger in PVI Group
  Arms: PVI Guided Fluid Therapy
Diagnostic Test: CVP Guided Fluid management during surgery for CVP<10 cms H2O colloid bolus will be given — Placement of central venous catheter
  Arms: CVP Guided Fluid Therapy

SUMMARY:
During major surgeries optimal intravenous fluid administration is essential , conventional method may cause fluid overload , increased extravascular Lung water can lead to postoperative cardio-respiratory complications , this study was designed to detect immediate postoperative EVLW with Lung Ultrasonography in patients receiving Central venous pressure Guided and Pleth variability Index (PVI) guided fluids intraoperatively .

DETAILED DESCRIPTION:
Standard General Anaesthesia with Endotracheal Tube and Intermittent Positive Pressure Ventilation (IPPV) was given to all patients,Monitoring included 5 lead ECG, Oxygen Saturation (SPO2), End tidal Carbon di oxide (ETCO2), Invasive Blood Pressure (IBP) , Central venous Pressure (CVP), Pleth variability Index (PVI) in study group and Bispectral Index (BIS) , Core temperature .Postintubation before commencement of surgery baseline Lung Ultrasonography will be performed with non-linear probe in 4 zones on Right and Left Lung-- Zone I Right Midclavicular in second intercostal space , Zone II Right Parasternal in third intercostal space, Zone III Anterior axillary line in fourth intercostal space Zone IV Posterior axillary line in the V intercostal space. Zone V to VIII in Corresponding spaces on the Left side . In the control Group CVP Guided IV fluids were given during surgery CVP will be maintained between 10-16 cms H20 , for CVP values < 10 cms H20 colloid bolus 200ml was given.In the Study Group PVI guided IV Fluids will be given to maintain PVI <12 for increase in PVI value > 12 Colloid bolus 200 ml will be given. After the completion of surgery and before extubation Lung Ultrasonography will be performed in all 8 Zones in both lungs to identify B Lines and total number of B lines will be calculated , Extra Vascular Lung Water (EVLW) Grading will be done as B Lines <5 Mild, between 5-15 moderate , > 15 severe .Total IV Fluids along with colloid boluses will be calculated , Postintubation as Baseline and after the completion of surgery Arterial blood gas analysis will be done for Alveolar-Arterial Oxygenation Pa02 (A-a) and blood Lactate values . After completion of surgery neuromuscular blockade will be reversed and trachea extubated .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major Oncosurgeries under General Anaesthesia

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF )< 40%
* Chronic Obstructive Pulmonary Disease (COPD)
* BMI >30
* Lung fibrosis
* Previous lung surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Extravascular Lung Water detection | End of surgery upto 1 hour
  At the end of surgery before extubation Lung Ultrasonography will be performed in 4 Zones bilaterally to detect total number of B lines in both groups

SECONDARY OUTCOMES:
Adequacy of Perfusion | End of surgery upto 1 hour
  Serum Blood Lactate levels will be measured at end of surgery in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anita C Kulkarni, MD, Principal Investigator — Rajiv Gandhi Cancer Institute and Research Centre
Locations (1):
- Rajiv Gandhi Cancer Institute and Research Centre, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Picano E, Pellikka PA. Ultrasound of extravascular lung water: a new standard for pulmonary congestion. Eur Heart J. 2016 Jul 14;37(27):2097-104. doi: 10.1093/eurheartj/ehw164. Epub 2016 May 12. PMID 27174289
- [Background] Anile A, Russo J, Castiglione G, Volpicelli G. A simplified lung ultrasound approach to detect increased extravascular lung water in critically ill patients. Crit Ultrasound J. 2017 Dec;9(1):13. doi: 10.1186/s13089-017-0068-x. Epub 2017 Jun 13. PMID 28612302